CLINICAL TRIAL: NCT02774161
Title: Quantitative Ultrasound Spectroscopy to Early HCC
Brief Title: B-mode Ultrasound Imaging in Detecting Early Liver Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Aya Kamaya, Professor of Radiology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-36299; NCI-2016-00663 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GIIMG0007 (Other: OnCore)
Record Dates: First submitted 2016-05-02; First posted 2016-05-17 (Estimated); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Cirrhosis; Early Hepatocellular Carcinoma; Fibrosis; Stage I Hepatocellular Carcinoma; Stage II Hepatocellular Carcinoma
MeSH Terms: conditions — Fibrosis; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (B-mode ultrasound imaging) (Experimental): Patients undergo B-mode ultrasound imaging of the liver over 15 minutes.
  Interventions: Other: Ultrasound Tomography

INTERVENTIONS:
Other: Ultrasound Tomography — Undergo B-mode ultrasound imaging

SUMMARY:
This pilot trial studies how well B-mode ultrasound imaging works in detecting liver cancer that is early in its growth and may not have spread to other parts of the body. Diagnostic procedures, such as B-mode ultrasound imaging, may help find and diagnose liver cancer and find out how far the disease has spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To investigate the use of quantitative ultrasound spectroscopy to detect early hepatocellular carcinoma (HCC) as an inexpensive and widely available quantitative (i.e. robust) method to confirm disease in developing countries.

OUTLINE:

Patients undergo B-mode ultrasound imaging of the liver over 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

For Healthy Volunteers

1. Patients over 18 years of age.
2. Must have no known medical problems and have had a full medical exam within 6 months of the study. If healthy volunteers have not had a full medical exam within 6 months of the study, one of the ultrasound physicians will conduct the medical exam prior to any study procedures.

For HCC patients

1. Patients over 18 years of age.
2. Patient with confirmed diagnosis of HCC, and untreated or Patients with Suspected HCC (Suspected HCC nodules should preferably be smaller than 3 cm and preferably within 6 cm in depth of the transducer head to minimize attenuation) and untreated or Patients at a higher risk of HCC undergoing a screening program by Ultrasound.

Exclusion Criteria:

For Healthy volunteers

1. Patients who are not likely to comply with the protocol requirements.

For HCC patients

1. Patients should not be taking other Investigational Agents.
2. Concomitant medications for treatment of the target lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-06-19 (Actual); Study Completion 2017-06-19 (Actual)

PRIMARY OUTCOMES:
Mid-band fit | Up to 16 months
  The Mid-band fit is related to the intensity of the returned ultrasound signal at different frequencies has been shown to change with tissue morphology.
Spectral intercept | Up to 16 months
  Spectral intercept (SI) is mostly related to the number scatterers and their density in the tissue. Changes in the SI have been demonstrated to occur due to different pathologies and result from treatments that change the structure of the tissue being imaged.
Spectral slope | Up to 16 months
  Summarized as the maximum and/or average value over the lesion of interest (using a region of interest selection) and the liver image as a whole.

CONTACTS AND LOCATIONS:
Overall Officials: Aya Kamaya, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Palo Alto, California, United States